CLINICAL TRIAL: NCT07222202
Title: A Noninvasive, Flexible Conductive Hearing Aid With Micro-epidermal Actuators on Pediatric and Adult Patients
Brief Title: Evaluation of Flexible Conductive Hearing Aids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00133858
Record Dates: First submitted 2025-10-28; First posted 2025-10-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Conductive Hearing Loss
Keywords: hearing aids; hearing loss
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss

STUDY DESIGN:
Intervention Model Description: Patients with conductive/mixed hearing loss will be assessed to observe their hearing threshold before using the hearing aid and reassessed with our hearing aid attached. Healthy subjects will wear noise-cancelling headphones and ear plugs to simulate conductive hearing loss, and their hearing threshold will be assessed before and during the flexible hearing aid attachment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- flexible Band-Aid style hearing device (Experimental): Patients with conductive/mixed hearing loss will be assessed to observe their hearing threshold before using the hearing aid and reassessed with our hearing aid attached. Healthy subjects will wear noise-cancelling headphones and ear plugs to simulate conductive hearing loss, and their hearing threshold will be assessed before and during the flexible hearing aid attachment.
  Interventions: Device: flexible conductive hearing aid

INTERVENTIONS:
Device: flexible conductive hearing aid — Eligible patients will wear hearing aids on flexible substrate and MEA (Micro epidermal actuator is a flexible material (e.g., plastics) to be placed on epidermis layer of skin for generating vibrations) on skull behind the ear or forehead. A neonatal adhesive, tape, Band-Aid or a headband will secure the aid/MEA on the skin.

SUMMARY:
Conductive hearing loss (CHL) is the most common type of hearing loss among the pediatric population. CHL occurs when sound is not properly transmitted from the external ear to the cochlea, and congenital pathologies like microtia/anotia, atresia, and absent or malformed ossicles make hearing loss permanent.

DETAILED DESCRIPTION:
Standard treatment for permanent conductive hearing loss includes osseointegrated implants, which require surgery and are invasive for pediatric patients. Conductive hearing loss can also be treated by non-surgical solutions such as wearable and behind-the-ear aids; however, they present challenges such as instability, stigmatization, and discomfort because of the device's design. Therefore, patients (ages 6 months to 80 years) with permanent (CHL) can benefit from a flexible, Band-Aid like hearing aid.

ELIGIBILITY:
Inclusion Criteria:

* Male and female infants, children, adolescents, and adult patients who are diagnosed with unilateral or bilateral mixed or conductive hearing loss
* Male and female patients seen at Atrium Health-Audiology for a clinical, standard of care office visit who have a diagnosis of conductive or mixed hearing loss and may currently wear hearing aids
* Male and female infants, children, adolescents, and adults who are candidates for conductive hearing aids (Osseo-integrated or wearable aids) or for canalplasty or ossicular chain reconstruction surgery
* Healthy subjects will include male and female infants, children, adolescents, and adults who do not have conductive or mixed hearing loss
* Pregnant women -are eligible for this study. Standard of Care allows pregnant patients to be fit for hearing aids without risk.

Exclusion Criteria:

* Adult patients unable to independently understand the purpose of the study and the procedures and/or who are not willing to participate

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Does the subject indicate hearing or states they can hear sound | Hour 1
  Voltage (with a maximum of 20 V, frequency range: 20 Hz to 20 kHz) will be applied to Micro epidermal actuator (MEA) through external power supply/function generator, or through amplifier in the hearing aid circuit. While wearing the device, they are asked to respond or repeat when they hear sound either delivered through the device or through the speaker on the wall in front of them. All sounds are presented at a comfortable level.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Moghimi, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participants data, collected during the trial after deidentification
Supporting Information: Study Protocol
Time Frame: Immediately after publication. No end date
Access Criteria: Any purposes